CLINICAL TRIAL: NCT03122652
Title: Multi-center, Randomized, Double-blinded Study of Teriflunomide® in Radiologically Isolated Syndrome (RIS) The TERIS Study
Brief Title: Randomized, Double-blinded Study of Treatment:Teriflunomide, in Radiologically Isolated Syndrome
Acronym: TERIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-PP-11
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: Radiologically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terifunomide (Experimental)
  Interventions: Drug: Teriflunomide 14 MG Oral Tablet [Aubagio]
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Teriflunomide 14 MG Oral Tablet [Aubagio] — 1 tablet once a day
  Arms: Terifunomide
Drug: Placebo Oral Tablet — 1 tablet once a day
  Arms: Placebo

SUMMARY:
Multiple sclerosis (MS) is a common cause of severe neurological disability in young adults, resulting from an autoimmune interruption of both myelin and axons within the central nervous system (CNS). The diagnosis is made by fulfilling both spatial criteria, by meeting the requisite number of lesions within the brain or spinal cord, along with criteria for time, by demonstrating a history of at least a second clinical attack or the development of a new MS lesion on MRI after the seminal neurological event. In the case of MS, healthy individuals who do not exhibit signs of neurological dysfunction commonly have brain MRI studies performed for a reason other than an evaluation for MS that reveal unexpected anomalies highly suggestive of demyelinating plaques given their size, location, and morphology. These healthy subjects lack symptomatology suggestive of MS and fulfill formal criteria for radiologically isolated syndrome (RIS), a recently described MS subtype that expands upon the phenotype of at-risk individuals for future demyelinating events. The discovery of such anomalies creates intersecting neuro-ethical, legal, social, and practical medical management quandaries and is, therefore, of both immediate and long-term clinical significance. Despite advancements in the characterization of RIS subjects, and in our understanding of risk factors for initial symptom development, the effect of treatment on such cases remain unclear.

The purpose of this investigation is to systematically study the efficacy of Teriflunomide in those individuals who possess incidental white matter anomalies within the brain and following a MRI study that is performed for a reason other than for the evaluation of MS.

RIS subjects are frequently exposed to disease modifying therapies despite the lack of scientific literature supporting the use of such treatments. Earlier treatment intervention may extend the time to the first acute or progressive clinical event resulting from CNS demyelination and reduce radiological progression. In addition, early treatment may result in more profound effects on reducing disability progression long-term.

The primary outcome measure for this trial is the time to the first acute or progressive neurological event resulting from CNS demyelination.

This study will include RIS subjects from the Europe who fulfill 2009 RIS Criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of all ages(>18 years and <65 years) meeting 2009 RIS criteria:

   A. The presence of incidentally identified CNS white matter anomalies meeting the following MRI criteria:
   1. Ovoid, well-circumscribed, and homogeneous foci observed with or without involvement of the corpus callosum
   2. T2 hyperintensities measuring ≥3 mm and fulfilling Barkhof criteria (at least three out of four) for dissemination in space
   3. Anomalies not following a clear vascular pattern
   4. Structural neuroimaging abnormalities identified not explained by another disease process B. No historical accounts of remitting clinical symptoms consistent with neurological dysfunction C. The MRI anomalies do not account for clinically apparent impairments in social, occupational, or generalized area of functioning D. The MRI anomalies are not due to the direct physiological effects of substances (recreational drug use, toxic exposure) or a medical condition E. Exclusion of individuals with MRI phenotypes suggestive of leukoaraiosis or extensive white matter changes lacking clear involvement of the corpus callosum F. The CNS MRI anomalies are not better accounted for by another disease process
2. Identified RIS cases with the initial MRI demonstrating anomalies suggestive of demyelinating disease dated ≥ 2009
3. Incidental anomalies identified on MRI of the brain or spinal cord with the primary reason for the acquired MRI resulting from an evaluation of a process other than MS
4. Affiliation to the social security system
5. Subjects of reproductive potential are eligible only if the following applies:

   * Women of childbearing potential (WOCBP):Must have a negative serum pregnancy test at Visit 1 (Screening) and negative urine pregnancy test at Visit 2 (Baseline);
   * Must be agree to undertake 1 monthly urine pregnancy tests during the study and up to 6 weeks after the first of two tests showing teriflunomide plasma level <0.02 mg/L;
   * Must agree to use reliable methods of contraception from Visit 1 until 6 weeks after the first oft wo tests showing teriflunomide plasma level <0.02 mg/L.

Fertile male subjects participating in the study who are sexually active with WOCBP:

- Must agree to use condom during the treatment period and for an additional 6 weeks after the first oft wo tests showing teriflunomide plasma level <0.02 mg/L.

Exclusion Criteria:

1. Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of summary of product characteristics (SmPC).
2. Patients with severe hepatic impairment (Child-Pugh class C).
3. Patients with severe immunodeficiency states, e.g. AIDS.
4. Patients with significantly impaired bone marrow function or significant anaemia, leucopenia, neutropenia or thrombocytopenia.
5. Patients with severe active infection until resolution.
6. Patients with severe renal impairment undergoing dialysis.
7. Patients with severe hypoproteinaemia, e.g. in nephrotic syndrome.
8. Lactating or pregnant women
9. Subjects wishing to parent a child during the study
10. Incomplete medical history or radiological data
11. History of remitting clinical symptoms consistent with multiple sclerosis lasting > 24 hours prior to CNS imaging revealing anomalies suggestive of MS
12. History of paroxysmal symptoms associated with MS (i.e. Lhermitte's or Uhthoff's phenomena)
13. CNS MRI anomalies are better accounted for by another disease process
14. The subject is unwilling or unable to comply with the requirements of the study protocol
15. Exposure to a disease modifying therapy within the past 3 months
16. Exposure to high-dose glucocorticosteroid treatment within the past 30 days
17. Vulnerable subject (such as deprived from freedom) as defined in Section 1.61 of International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP: Individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples are members of a group with a hierarchical structure, such as medical, pharmacy, dental, and nursing students, subordinate hospital and laboratory personnel, employees of the pharmaceutical industry, members of the armed forces, and persons kept in detention. Other vulnerable subjects include patients with incurable diseases, persons in nursing homes, unemployed or impoverished persons, patients in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, minors, and those incapable of giving consent.)
18. Participation in another clinical trial of an investigational medicinal product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Time to the first acute or progressive neurological event resulting from CNS demyelination. | Week 96
  Acute neurological event: The development of an acute neurological episode localized to the optic nerve, brainstem, cerebellum, spinal cord, or long sensory or motor tracts, lasting > 24 hours followed by a period of symptom improvement.
  Progressive event: The onset of a clinical symptom (e.g. leg weakness) with the temporal profile revealing at least a 12-month progression of neurological deficits.

SECONDARY OUTCOMES:
New or enlarging T2 lesions | Week 48
  Number of new or enlarging T2 lesions on MRI
New or enlarging T2 lesions | Week 96
  Number of new or enlarging T2 lesions on MRI
New contrast enhancing lesions | Week 48
  New contrast enhancing lesions on MRI
New contrast enhancing lesions | Week 96
  New contrast enhancing lesions on MRI
New T2-lesion volumes | Week 48
  New T2-lesion volumes on MRI
New T2-lesion volumes | Week 96
  New T2-lesion volumes on MRI
Brain atrophy | Week 96
  Brain atrophy on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Christine LEBRUN-FRENAY, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (23):
- France (15):
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHRU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - APHP - Hôpital La Pitié Salpêtrière, Paris
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
- Inselspital Bern, Bern, Switzerland
- Turkey (Türkiye) (7):
  - Hacettepe University, Ankara
  - Mustafa Kemal University, Antakya
  - Uludag University School of Medicine, Bursa
  - Istanbul University, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli University School of Medicine, Kocaeli
  - Ondokuz Mayis University, Faculty of Medicine, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lebrun-Frenay C, Siva A, Sormani MP, Landes-Chateau C, Mondot L, Bovis F, Vermersch P, Papeix C, Thouvenot E, Labauge P, Durand-Dubief F, Efendi H, Le Page E, Terzi M, Derache N, Bourre B, Hoepner R, Karabudak R, De Seze J, Ciron J, Clavelou P, Wiertlewski S, Turan OF, Yucear N, Cohen M, Azevedo C, Kantarci OH, Okuda DT, Pelletier D; TERIS Study Group. Teriflunomide and Time to Clinical Multiple Sclerosis in Patients With Radiologically Isolated Syndrome: The TERIS Randomized Clinical Trial. JAMA Neurol. 2023 Oct 1;80(10):1080-1088. doi: 10.1001/jamaneurol.2023.2815. PMID 37603328